CLINICAL TRIAL: NCT01871285
Title: An Evaluation of the Tolerability of Switching Subjects on Chronic Around-the-Clock (ATC) Opioid Therapy to Buprenorphine HCl Buccal Film
Brief Title: Evaluation of the Tolerability of Switching Subjects on Chronic ATC Opioid Therapy to Buprenorphine HCl Buccal Film
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: EN3409-204
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Pain
Keywords: ATC, Opioid, withdrawal, switch
MeSH Terms: conditions — Pain; Ataxia Telangiectasia | interventions — Buprenorphine; Oxycodone; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MSE Dose Group 1 (Experimental): Morning and evening dose of buprenorphine HCl buccal film (300 μg) + placebo capsule in one period, and then placebo film + over-encapsulated ATC opioid (morphine sulfate or oxycodone) at 50% MSE daily dose in the alternate period
  Interventions: Drug: Buprenorphine; Drug: Placebo film; Drug: Oxycodone; Drug: Morphine sulfate; Drug: Placebo capsule
- MSE Dose Group 2 (Experimental): Morning and evening dose of buprenorphine HCl buccal film (450 μg) + placebo capsule in one period, and then placebo film + over-encapsulated ATC opioid (morphine sulfate or oxycodone) at 50% MSE daily dose in the alternate period
  Interventions: Drug: Buprenorphine; Drug: Placebo film; Drug: Oxycodone; Drug: Morphine sulfate; Drug: Placebo capsule

INTERVENTIONS:
Drug: Buprenorphine
  Other Names: Buprenorphine buccal film; Buprenorphine HCl buccal film; EN3409; BEMA Buprenorphine; BELBUCA
Drug: Placebo film — Matching placebo buccal film
  Other Names: Placebo buccal film; BEMA placebo
Drug: Oxycodone — Oxycodone extended-release (ER) or immediate-release (IR) 5, 10, 15, 20, and 30 mg over-encapsulated oral tablets
  Other Names: Oxycodone tablets; OxyContin; Oxycodone IR
Drug: Morphine sulfate — Morphine sulfate 15, 30, and 60 mg ER or 15 and 30 mg IR over-encapsulated oral tablets
  Other Names: Morphine sulfate tablets; MS Contin; Morphine sulfate IR
Drug: Placebo capsule — Oral placebo capsules matching the over-encapsulated morphine sulfate and oxycodone tablets
  Other Names: Matching placebo capsules

SUMMARY:
The primary aim of this study is to determine if chronic pain subjects on around-the-clock opioids who are receiving 100 to 220 mg oral morphine sulfate equivalent (MSE) can be safely transitioned on to buprenorphine hydrochloride (HCl) buccal film at 50% of their MSE dose without inducing opioid withdrawal or reversing analgesic effects.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-related procedure being performed
2. Male or non-lactating female subjects 18 to 60 years of age at time of consent
3. Female subjects who are non-pregnant on the basis of screening serum pregnancy test and who are practicing abstinence or using a medically acceptable form of contraception (eg, intrauterine device, hormonal birth control, or double barrier method) or have been post-menopausal, biologically sterile, or surgically sterile (ie, hysterectomy, bilateral oophorectomy, or tubal ligation) for more than 1 year
4. Male subjects who are practicing abstinence, surgically sterile or are using a medically acceptable form of contraception
5. Subjects with a ≥6 months history of chronic pain (including peripheral neuropathic pain) requiring ATC opioid therapy with ≥80 mg but ≤220 mg MSE per day for at least 28 days
6. Receiving one of the following opioids ATC for ≥28 days: (i) Morphine Sulfate; (ii) Oxycodone hydrochloride
7. Displays signs and symptoms of withdrawal (ie, COWS score ≥5) within 5 minutes following naloxone challenge
8. Able to understand the study procedures, complete the assessment scales, and communicate meaningfully with study personnel
9. Stable health, as determined by the Principal Investigator, on the basis of medical history, physical examination, and screening laboratory results

Exclusion Criteria:

1. Inability to meet study participation requirements, including two 2-night stays with pharmacokinetic sampling
2. A history or current evidence of clinically significant pulmonary (eg, asthma, chronic obstructive pulmonary disease, cor pulmonale or severe bronchial asthma ), gastrointestinal, hepatic, renal, hematologic, immunologic, endocrine, neurologic, oncologic or psychiatric disorder or any other condition, including evidence of abnormalities on physical examination, abnormal vital signs, electrocardiogram (ECG), or clinical laboratory values which in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results
3. Supine systolic blood pressure >180 mm Hg or <90 mm Hg or diastolic blood pressure > 105 mm Hg or <50 mm Hg at screening (may be repeated once)
4. COWS score greater than 4 prior to the screening naloxone challenge
5. Aspartate aminotransferase or alanine aminotransferase >3 times the upper limits of normal or serum creatinine >1.9 mg/dL at Screening, or any laboratory abnormality which, in the opinion of the Investigator, would contraindicate study participation
6. Use of monoamine oxidase inhibitors within 14 days of screening or during the study
7. Use of any medication, nutraceutical or herbal product with cytochrome P450 3A4 inhibition or induction properties within the past 30 days
8. Donation of 450 mL or more of blood within 30 days prior to screening or a hemoglobin value <11.0 g/dL at screening
9. Documented history of alcohol and/or substance abuse (excluding nicotine and/or caffeine) within 5 years prior to screening, and/or is currently in treatment or is seeking treatment for alcohol and/or substance abuse, as assessed by the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) criteria
10. Positive alcohol breath test at screening
11. Positive urine toxicology screen for drugs of abuse at screening
12. History of hypersensitivity, allergy, or contraindication to any opioid or clinically significant intolerance to buprenorphine or naloxone
13. History of seizures, convulsions, or increased intra-cranial pressure (history of pediatric febrile seizures is permitted)
14. History of significant head injury within 6 months of screening
15. Any clinically significant abnormality of the buccal mucosa which could impact drug absorption
16. Participation in the treatment phase of a clinical research study involving any investigational drug within 28 days (or 5 elimination half-lives, whichever is longer) of screening
17. Previous participation in this clinical study or any other clinical study involving BEMA buprenorphine (buprenorphine HCl buccal film)
18. In the Investigator's opinion at significant risk for suicidal behavior based on the Columbia Suicide Severity Rating Scale (C-SSRS)
19. Hypokalemia or clinically unstable cardiac disease, including unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, or active myocardial ischemia
20. History of myocardial infarction
21. Corrected QT interval (QTcF) of ≥450 milliseconds on the 12-lead ECG
22. History of long QT syndrome or a family member with this condition
23. Use of class IA antiarrhythmic medications or class III antiarrhythmic medications within 14 days of screening
24. Current use of α2 agonist antihypertensives (eg, clonidine), 5-HT3 antagonists (eg, ondansetron), benzodiazepines, or other medications that would be anticipated to confound detection of signs and symptoms of opioid withdrawal
25. Involvement in the planning and/or conduct of the study (applies to both sponsor or designee staff and staff at the study sites)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Kirby, PhD, Study Director — Endo Pharmaceuticals
Locations (3):
- United States (3):
  - Vince and Associates Clinical Research, Inc., Overland Park, Kansas
  - CRI Lifetree, Philadelphia, Pennsylvania
  - CRI Lifetree (Lifetree Clinical Research), Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with at least 6 months history of chronic pain requiring around-the-clock (ATC) opioid therapy with 80 to 220 mg morphine sulfate equivalent (MSE) per day for at least 28 days
Pre-assignment Details: Subjects were enrolled and entered a screening period (73). Those meeting criteria for study entry including positive precipitated withdrawal during naloxone challenge (39) were randomized and stratified to 2 dose groups (subjects requiring 80-160 mg MSE/day ATC to MSE Dose Group 1 and subjects requiring 161-220 mg MSE/day ATC to MSE Dose Group 2).
Groups:
- MSE Dose Group 1 (AB) - Buprenorphine (300 μg) Then ATC Opioid: MSE Dose Group 1 receiving treatment sequence AB with A being buprenorphine hydrochloride (HCl) buccal film (300 μg) + placebo ATC morning and evening in period 1 and B being ATC opioid + placebo buccal film morning and evening in period 2. Each period included 1 treatment day.
- MSE Dose Group 1 (BA) - ATC Opioid Then Buprenorphine (300 μg): MSE Dose Group 1 receiving treatment sequence BA with B being ATC opioid + placebo buccal film morning and evening in period 1 and A being buprenorphine HCl buccal film (300 μg) + placebo ATC morning and evening in period 2. Each period included 1 treatment day.
- MSE Dose Group 2 (AB) - Buprenorphine (450 μg) Then ATC Opioid: MSE Dose Group 2 receiving treatment sequence AB with A being buprenorphine HCl buccal film (450 μg) + placebo ATC morning and evening in period 1 and B being ATC opioid + placebo buccal film morning and evening in period 2. Each period included 1 treatment day.
- MSE Dose Group 2 (BA) - ATC Opioid Then Buprenorphine (450 μg): MSE Dose Group 2 receiving treatment sequence BA with B being ATC opioid + placebo buccal film morning and evening in period 1 and A being buprenorphine HCl buccal film (300 μg) + placebo ATC morning and evening in period 2. Each period included 1 treatment day.
Period: First Intervention (1 Day)
Arm/Group | MSE Dose Group 1 (AB) - Buprenorphine (300 μg) Then ATC Opioid | MSE Dose Group 1 (BA) - ATC Opioid Then Buprenorphine (300 μg) | MSE Dose Group 2 (AB) - Buprenorphine (450 μg) Then ATC Opioid | MSE Dose Group 2 (BA) - ATC Opioid Then Buprenorphine (450 μg)
Started | 18 | 15 | 4 | 2
Completed | 17 | 14 | 3 | 2
Not Completed | 1 | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Period: Second Intervention (1 Day)
Arm/Group | MSE Dose Group 1 (AB) - Buprenorphine (300 μg) Then ATC Opioid | MSE Dose Group 1 (BA) - ATC Opioid Then Buprenorphine (300 μg) | MSE Dose Group 2 (AB) - Buprenorphine (450 μg) Then ATC Opioid | MSE Dose Group 2 (BA) - ATC Opioid Then Buprenorphine (450 μg)
Started | 17 | 14 | 3 | 2
Completed | 17 | 14 | 3 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis is based on Safety population; all subjects who received at least 1 dose of double-blind double dummy treatment.
Groups:
- MSE Dose Group 1: Morning and evening dose of buprenorphine HCl buccal film (300 μg) + placebo capsule in one period, and then placebo buccal film + over-encapsulated ATC opioid at 50% MSE daily dose in the alternate period
- MSE Dose Group 2: Morning and evening dose of buprenorphine HCl buccal film (450 μg) + placebo capsule in one period, and then placebo buccal film + over-encapsulated ATC opioid at 50% MSE daily dose in the alternate period
- Total: Total of all reporting groups
Arm/Group | MSE Dose Group 1 | MSE Dose Group 2 | Total
Number analyzed (Participants) | 33 | 6 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 6 | 39
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 43.0 [26 to 55] | 44.0 [31 to 60] | 43.0 [26 to 60]
Gender [Count of Participants; unit: Participants]
  Female | 17 | 4 | 21
  Male | 16 | 2 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders
Description: A responder is defined as a subject whose maximum (across all time points) clinical opiate withdrawal scale (COWS) total score is ≥13. COWS scores range 0 to 4 or 5 on 11 items related to opiate withdrawal signs or symptoms; total score range 0 to 48 where 0-4 = no withdrawal and 5-12 = mild, 13-24 = moderate, 25-36 = moderately severe, more than 36 = severe withdrawal.
Time Frame: Pre-dose (-0.5), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 9, 12, 12.5, 13, 13.5, 14, 16, and 24 (or end of study visit) hours post 1st study drug dose on each day of administration (period 1 [day 1] and period 2 [day 2]) in each treatment sequence
Population: Analysis based on Per-protocol population (all randomized subjects who did not have major protocol deviations that might have confounded interpretation of the COWS [eg, received erroneous treatment], completed both crossover periods, and provided at least the first 4 hours of COWS data for each of the 2 treatment periods); 4 subjects were excluded.
Measure: Number; unit: participants
Groups:
- MSE Dose Group 1 - Buprenorphine: Subjects requiring 80-160 mg MSE per day (ATC) received 2 doses of buprenorphine HCl buccal film (300 μg) and 2 doses of ATC opioid at 50% MSE total daily dose (TDD); following exposure to buprenorphine
- MSE Dose Group 1 - ATC Opioid: Subjects requiring 80-160 mg MSE per day (ATC) received 2 doses of buprenorphine HCl buccal film (300 μg) and 2 doses of ATC opioid at 50% MSE TDD; following exposure to ATC opioid
- MSE Dose Group 2 - Buprenorphine: Subjects requiring 161-220 mg MSE per day (ATC) received 2 doses of buprenorphine HCl buccal film (450 μg) and 2 doses of ATC opioid at 50% MSE TDD; following exposure to buprenorphine
- MSE Dose Group 2 - ATC Opioid: Subjects requiring 161-220 mg MSE per day (ATC) received 2 doses of buprenorphine HCl buccal film (450 μg) and 2 doses of ATC opioid at 50% MSE TDD; following exposure to ATC opioid
Arm/Group | MSE Dose Group 1 - Buprenorphine | MSE Dose Group 1 - ATC Opioid | MSE Dose Group 2 - Buprenorphine | MSE Dose Group 2 - ATC Opioid
Number analyzed (Participants) | 31 | 31 | 4 | 4
participants | 1 | 2 | 0 | 0

2. Secondary Outcome: Change From Baseline in COWS Total Score Over Time
Description: Investigator-rated COWS scores range 0 to 4 or 5 on 11 items related to opiate withdrawal signs or symptoms; total score range 0 to 48 where 0-4 = no withdrawal and 5-12 = mild, 13-24 = moderate, 25-36 = moderately severe, more than 36 = severe withdrawal.
Time Frame: Pre-dose (-0.5; baseline), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 9, 12, 12.5, 13, 13.5, 14, 16, and 24 (or end of study visit) hours post 1st study drug dose on each day of administration (period 1 [day 1] and period 2 [day 2]) in each treatment sequence
Population: Analysis based on Per-protocol population (all randomized subjects who did not have major protocol deviations that might have confounded interpretation of the COWS [eg, received erroneous treatment], completed both crossover periods, and provided at least the first 4 hours of COWS data for each of 2 treatment periods); 4 subjects were excluded.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | MSE Dose Group 1 - Buprenorphine | MSE Dose Group 1 - ATC Opioid | MSE Dose Group 2 - Buprenorphine | MSE Dose Group 2 - ATC Opioid
Number analyzed (Participants) | 31 | 31 | 4 | 4
score
  Hour 0.5 | 0.1 (0.67) | -0.3 (1.47) | 0.0 (0.82) | -1.3 (0.96)
  Hour 1 | 0.3 (1.04) | 0.0 (1.94) | 0.8 (1.50) | -1.0 (1.41)
  Hour 1.5 | 0.4 (1.31) | 0.2 (2.50) | 0.5 (1.29) | -1.0 (1.41)
  Hour 2 | 0.3 (0.90) | 0.2 (2.48) | 1.8 (1.50) | -1.0 (0.82)
  Hour 2.5 | 0.6 (1.41) | 0.3 (2.32) | 1.3 (1.26) | -1.0 (0.82)
  Hour 3 | 0.6 (1.72) | 0.2 (2.49) | 0.3 (0.96) | -1.0 (1.63)
  Hour 3.5 | 0.9 (1.81) | 0.3 (2.17) | 1.5 (1.73) | -0.8 (1.71)
  Hour 4 | 0.8 (1.54) | 0.4 (2.48) | 1.0 (1.15) | -1.0 (1.83)
  Hour 6 | 0.6 (1.58) | 0.6 (2.76) | 1.0 (1.15) | 0.0 (2.58)
  Hour 9 | 0.9 (1.47) | 1.4 (3.64) | 1.3 (1.26) | 1.0 (1.15)
  Hour 12 | 2.1 (2.38) | 1.5 (3.43) | 3.3 (2.50) | 0.3 (3.77)
  Hour 12.5 | 1.0 (1.32) | 0.5 (2.01) | 3.0 (3.56) | 1.3 (4.27)
  Hour 13 | 0.9 (1.26) | 0.5 (1.72) | 3.3 (3.77) | 0.0 (3.83)
  Hour 13.5 | 1.0 (1.76) | 0.4 (1.80) | 1.8 (2.63) | -0.3 (3.40)
  Hour 14 | 0.7 (1.33) | 0.2 (2.06) | 3.3 (3.10) | -0.3 (3.10)
  Hour 16 | 0.5 (1.55) | -0.1 (1.88) | 1.8 (2.06) | -0.3 (3.10)
  Hour 24 | 1.8 (3.13) | 0.7 (3.12) | 2.0 (2.58) | 2.8 (2.63)

3. Secondary Outcome: Change From Baseline in "Pain Now" Over Time Using NRS
Description: Subject rating of pain intensity using 11-point numerical rating scale (NRS) where 0=no pain and 10=pain as bad as you can imagine.
Time Frame: Pre-dose (-0.5; baseline), 0.5, 1, 2, 4, 9, 12, 12.5, 13, 14, 16, and 24 (or end of study visit) hours post 1st study drug dose on each day of administration (period 1 [day 1] and period 2 [day 2]) in each treatment sequence
Population: Analysis based on Per-protocol population (all randomized subjects who did not have major protocol deviations that might have confounded interpretation of the COWS [eg, received erroneous treatment], completed both crossover periods, and provided at least the first 4 hours of COWS data for each of the 2 treatment periods); 4 subjects excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MSE Dose Group 1 - Buprenorphine | MSE Dose Group 1 - ATC Opioid | MSE Dose Group 2 - Buprenorphine | MSE Dose Group 2 - ATC Opioid
Number analyzed (Participants) | 31 | 31 | 4 | 4
units on a scale
  Hour 0.5 | -0.3 (1.24) | -0.6 (0.92) | -0.5 (1.73) | -1.3 (0.50)
  Hour 1 | -0.5 (1.43) | -1.1 (1.30) | 0.3 (1.26) | -1.5 (1.00)
  Hour 2 | -0.7 (1.37) | -1.2 (1.49) | 0.8 (0.96) | -1.3 (1.50)
  Hour 4 | -0.9 (1.97) | -1.0 (1.80) | 0.5 (1.73) | -1.8 (2.06)
  Hour 9 | -0.5 (2.29) | -0.1 (1.97) | 1.0 (1.41) | -0.8 (2.06)
  Hour 12 | 0.5 (2.13) | 0.3 (2.01) | 1.5 (1.91) | -0.3 (2.63)
  Hour 12.5 | 0.0 (2.29) | -0.4 (2.01) | 1.0 (2.16) | -0.3 (2.99)
  Hour 13 | -0.4 (2.40) | -0.7 (2.07) | 0.8 (1.89) | -0.8 (2.99)
  Hour 14 | -0.7 (2.24) | -1.2 (2.02) | 1.0 (2.16) | -1.0 (3.37)
  Hour 16 | -0.9 (2.37) | -1.4 (2.03) | 0.3 (2.22) | -1.3 (3.30)
  Hour 24 | -0.2 (2.45) | -0.2 (2.12) | 0.8 (2.99) | 0.0 (2.94)

4. Primary Outcome: Maximum COWS Total Score
Description: Investigator-rated COWS scores range 0 to 4 or 5 on 11 items related to opiate withdrawal signs or symptoms; total score range 0 to 48 where 0-4 = no withdrawal and 5-12 = mild, 13-24 = moderate, 25-36 = moderately severe, more than 36 = severe withdrawal. The maximum COWs total score is defined as the maximum COWs total score across all time points during the corresponding treatment period after study drug administration for each subject.
Time Frame: as for outcome 1
Population: Analysis based on Per-protocol population (all randomized subjects who did not have major protocol deviations that might have confounded interpretation of the COWS [eg, received erroneous treatment], completed both crossover periods, and provided at least the first 4 hours of COWS data for each of 2 periods); 4 subjects were excluded.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | MSE Dose Group 1 - Buprenorphine | MSE Dose Group 1 - ATC Opioid | MSE Dose Group 2 - Buprenorphine | MSE Dose Group 2 - ATC Opioid
Number analyzed (Participants) | 31 | 31 | 4 | 4
score | 4.6 (3.15) | 5.3 (4.42) | 5.5 (1.91) | 6.3 (2.50)
Statistical Analysis 1: Comparison: MSE Dose Group 1 - Buprenorphine vs MSE Dose Group 1 - ATC Opioid; Test type: Superiority or Other; p = .7942, Mixed Models Analysis; Mean Difference (Final Values) = -0.182, 95% CI 2-sided [-1.60 to 1.24]
Statistical Analysis 2: Comparison: MSE Dose Group 2 - Buprenorphine vs MSE Dose Group 2 - ATC Opioid; Test type: Superiority or Other; p = .6155, Mixed Models Analysis; Mean Difference (Final Values) = 0.683, 95% CI 2-sided [-11.89 to 13.25]

5. Primary Outcome: Change From Baseline in Maximum COWS Total Score
Description: Investigator-rated COWS scores range 0 to 4 or 5 on 11 items related to opiate withdrawal signs or symptoms; total score range 0 to 48 where 0-4 = no withdrawal and 5-12 = mild, 13-24 = moderate, 25-36 = moderately severe, more than 36 = severe withdrawal. The change from baseline in maximum COWS total score is determined as the difference between the maximum COWs total score and the baseline COWs total score.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score
Arm/Group | MSE Dose Group 1 - Buprenorphine | MSE Dose Group 1 - ATC Opioid | MSE Dose Group 2 - Buprenorphine | MSE Dose Group 2 - ATC Opioid
Number analyzed (Participants) | 31 | 31 | 4 | 4
score | 4.0 (2.92) | 3.9 (4.11) | 4.5 (1.73) | 4.3 (1.89)
Statistical Analysis 1: Comparison: MSE Dose Group 1 - Buprenorphine vs MSE Dose Group 1 - ATC Opioid; Test type: Superiority or Other; p = .7942, Mixed Models Analysis; Mean Difference (Final Values) = -0.182, 95% CI 2-sided [-1.60 to 1.24]
Statistical Analysis 2: Comparison: MSE Dose Group 2 - Buprenorphine vs MSE Dose Group 2 - ATC Opioid; Test type: Superiority or Other; p = .6155, Mixed Models Analysis; Mean Difference (Final Values) = 0.683, 95% CI 2-sided [-11.89 to 13.25]

ADVERSE EVENTS:
Time Frame: From screening through follow-up contact 7-14 days after last dose (up to 7 weeks)
Description: Analysis based on Safety population; all subjects who received at least 1 dose of double-blind, double-dummy treatment
Groups:
- MSE Dose Group 1 - Buprenorphine: Subjects in MSE Dose Group 1 who received at least one 300-μg buprenorphine HCl buccal film in either period
- MSE Dose Group 1 - ATC Opioid: Subjects in MSE Dose Group 1 who received at least 1 dose of assigned ATC opioid in either period
- MSE Dose Group 2 - Buprenorphine: Subjects in MSE Dose Group 2 who received at least one 450-μg buprenorphine HCl buccal film in either period
- MSE Dose Group 2 - ATC Opioid: Subjects in MSE Dose Group 2 who received at least 1 dose of assigned ATC opioid in either period
Arm/Group | MSE Dose Group 1 - Buprenorphine | MSE Dose Group 1 - ATC Opioid | MSE Dose Group 2 - Buprenorphine | MSE Dose Group 2 - ATC Opioid
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/32 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 18/32 | 13/32 | 1/6 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MSE Dose Group 1 - Buprenorphine (N=32) | MSE Dose Group 1 - ATC Opioid (N=32) | MSE Dose Group 2 - Buprenorphine (N=6) | MSE Dose Group 2 - ATC Opioid (N=5)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MSE Dose Group 1 - Buprenorphine (N=32) | MSE Dose Group 1 - ATC Opioid (N=32) | MSE Dose Group 2 - Buprenorphine (N=6) | MSE Dose Group 2 - ATC Opioid (N=5)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 3 (3) | 4 (4) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (8) | 5 (5) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI and Institution reserve the right to publish and present the results of the work performed provided that Institution and/or PI submits a copy of any proposed publication to Sponsor's agent for review and comment at least 90 days in advance of its presentation or submission for publication. In addition, if Sponsor's agent requests, Institution and/or PI will withhold publication or presentation for an additional 60 days to allow for establishing and preserving its proprietary rights.